CLINICAL TRIAL: NCT04008472
Title: Telemedicine - Evaluation of the Impact of a Telemedicine Device (DTM) on the Prevention of Emergency Department Visits and Hospitalizations of Nursing Home Residents Aged Polypathological
Acronym: GERONTACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I14036 - GERONTACCESS
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-07

CONDITIONS: Polypathology
Keywords: Telemedecine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedecine (Experimental): Patients benefiting from telemedicine
  Interventions: Other: Telemedecine
- Control (No Intervention): routine care without telemedecine

INTERVENTIONS:
Other: Telemedecine — Initiation of tele-medical consultation with the resident, a caregiver for the nursing home, the referring physician and geriatrician téléexpert. After a overall geriatric assessment in nursing homes by UPSAV the first teleconsultation is organized within 10 days. Subsequent visits are scheduled every 3 months for 12 months. Spontaneous visits can be requested at the initiative of the referring physician.
  Arms: Telemedecine

SUMMARY:
For several decades, there is an aging population, particularly in industrialized countries. This lengthening of the duration of life is accompanied by an increase in the number of chronically ill patients. On an estimate of 15 million patients in France today, the figure reported for 2020 would be 20 million patients. Chronic diseases are responsible for functional decompensation and admission responsible autonomy breaks in nursing homes (Accommodation Establishment of People Dependent Elderly).

An estimated 700,000 the number of people currently living in retirement homes in France. These residents are mostly dependent and multiple pathologies requiring regular general and specialist medical monitoring . Medical concern demographic outlook and the need for access to quality care across the country leads to the development of telemedicine.

The need for telemedicine is not the same throughout the territory. It is less, or different, in highly urbanized areas where the density of health professionals is high, then it can be a new response to the needs of rural, isolated or landlocked. Telemedicine promotes the development of the concept of graduated care sector, especially in the management of patients with chronic diseases.

Telemedicine in rural nursing homes and can be a tool for assessing, monitoring and coordination to avoid decompensation of chronic conditions and rehospitalization.

This organization can afford to break the isolation of general practitioners and EHPAD coordinators physicians in rural areas and provide access to several specialties.

ELIGIBILITY:
Inclusion Criteria:

* Resident in one of 9 nursing homes participating in the project
* Resident polypathologique has at least two comorbidities
* Having made no request to change place of residence at the time of the inclusion visit
* Having given free consent, informed writing and signed by himself and / or his legal representative

Exclusion Criteria:

* Unaffiliated resident or non-receiving of social security
* severe pathology (ies) involving life-threatening in the short term
* Resident whose return home, transfer to another nursing home or to a long term care unit is programmed

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of telemedicine on prevention in old and polypathological patients | After 12 months
  Proportion of patients with emergency admission or unscheduled hospitalization in medical or surgical service over 12 months.

SECONDARY OUTCOMES:
Medico-economic impact | After 12 months
  cost effectiveness of the telemedicine device
Impact on recurring hospitalizations | After 12 months
  Number of readmissions
Impact on overall health | After 12 months
  Number of emergency admissions Number of readmissions Number of days of hospitalization Number of medical consultations o
Impact on the quality of life ( EQ5D questionnary) | After 12 months
  The EQ-5D (Europen Qyuality of llive) five dimension scale) questionnaire has two components: health state description and evaluation.
  In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are.
  Higher values represent a worse outcome.
  The scale ranges from 5 to 15.
Impact on mortality | After 12 months
  Proportion of patients who died at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Achille TCHALLA, Professor, Principal Investigator — University Hospital, Limoges